CLINICAL TRIAL: NCT06686264
Title: Effects of Core Stability Exercises on Motor Control in Patients With Low Back Pain.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Riphah IU Saman
Record Dates: First submitted 2024-11-12; First posted 2024-11-13 (Actual); Last update posted 2025-04-18 (Actual); Status verified 2025-04

CONDITIONS: Low Back Pain
Keywords: motor control; low back pain; core stability; motor control impairment
MeSH Terms: conditions — Low Back Pain

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Core stability Group A (Experimental): the core stability group includes core stability exercises along with the general back, pelvis and piriformis stretches
  Interventions: Other: core stability group A
- Traditional therapy group B (Active Comparator): the traditional group includes general back, pelvis and piriformis stretches
  Interventions: Other: traditional exercises group B

INTERVENTIONS:
Other: core stability group A — Abdominal hollowing in supine (10 reps & 2 sets) Single leg bridge (10 reps & 2 sets), 3 session per week for 6 weeks Prone Single leg raise(10 reps & 2 sets) Double leg bridge (10 reps & 2 sets) Abdominal hallowing in 4 point kneeling(10 reps & 2 sets), Complete Back stretch Pelvic rotations Posterior Pelvic tilt Knee to chest Piriformis stretch Maitland mobilization ( based on assessment) 10 reps 10 sec hold 2 session per day
  Arms: Core stability Group A
Other: traditional exercises group B — Complete Back stretch Pelvic rotations, 3 sessions per week for 6 week Posterior Pelvic tilt Knee to chest Piriformis stretch Maitland mobilization ( based on assessment) 10 reps 10 sec hold 2 session per day
  Arms: Traditional therapy group B

SUMMARY:
The aim of this research is aims to evaluate the effectiveness of core stability exercise on motor control, pain and disability in patients with low back pain.

Randomized controlled trials will be done at Rehman Medical Institute. The sample size was 44. The subjects were divided in two groups, 22 subjects were given conventional therapy and 22 were given conventional therapy along with core stability exercises. Study duration was of 6 months. Sampling technique applied was non probability convenience sampling technique. Patient with age 30-50 years both Male & female gender Presence of back pain for ≥6 weeks, MCI (Motor Control Impairment) complaints (pain provocation in static posture) with 3 or more positive tests were included. Tools used in the study are NPRS, ODI, and MCI tests.

DETAILED DESCRIPTION:
: Low back pain is a major health and socioeconomic problem and is associated with high costs in care, work absenteeism, and disability worldwide. According to evidence-based guidelines up to 90% of all Low Back Pain is classified as non-specific low back pain (NSLBP).Low back pain affects most people at some point in their lives, with up to an 84% lifetime prevalence and the prevalence depends on factors such as gender, age, educational level and occupation.

The underlying hypothesis is that impaired motor control (MC) and a lack of awareness of maladaptive movement patterns perpetuate Low Back Pain. Physiotherapists make clinical decisions based on the observation of movement control. O'Sullivan describes back pain patients with reduced Motor Control and excessive movement as pain provocateurs. Movement impairment syndromes and the detection of disordered movement, or pathokinesiology, is a key competence of physiotherapy. Pathokinesiologic movement patterns in the lumbar spine have been investigated and described, resulting in the publication of both reliability and validation studies of the examination procedures used. However, no clear evidence exists as to whether improvement in movement control can also lead to decreased pain and experienced daily disability in patients with NSLBP. Patients with Motor Control Impairment MCI present with mechanically induced pain in static postures together with visible movement abnormalities, such as decreased or increased movement of parts of the lumbar spine, or discrepancies in the proportion of hip, leg and spine movements. It is assumed that these movement abnormalities are influenced by current pain, previous pain episodes and the belief that pain provoked by movement is harmful. Patients exhibiting Motor Control Impairment demonstrate clinical features that can be screened with the aid of various clinical tests. Based on this principle, treatment aimed at restoring movement control, correcting movement patterns and avoiding pain-provoking postures could benefit patients with MCI.

The European Guidelines for Management of Chronic Non-Specific LBP recommend supervised exercise therapy as a first-line treatment for chronic Low Back Pain LBP. Exercise is the main treatment for chronic low back pain (CLBP) which is endorsed in most clinical practice guidelines. There is controversy over the most beneficial exercise, and there is little evidence that a particular kind of exercise is superior to another one.

In literature, there are studies which have been carried out for the effectiveness of exercises based on specific movement control findings in the low back, formed the justification for current study to evaluate core stability exercises in a subgroup of patients with non-specific LBP and impaired movement control or Motor control Impairment. Widely used synonyms for movement impairment syndromes are motor control dysfunctions and MC impairment. A study in Switzerland was carried out to observe improvement in Motor Control, decreased pain and disability in patients with NSLBP pain. The biggest effect was shown in the improvement of movement control ability following specific exercise intervention. A significant difference between patients with LBP and subjects without back pain regarding their ability to actively control the movements of the low back has been demonstrated in a study. One study was carried out to see the effects of movement control exercises versus general exercises on the disability and pain to patients with NSLBP and MCI but they both appeared equally effective in the patient subgroup included in this study After reviewing existing literature, it is notable that core stability exercises and other specific exercises have been frequently employed in studies focusing on the treatment of non-specific low back pain, yielding promising results in reducing pain and disability among patients. It is from evidence that patients with NSLBP exhibit Motor Control Impairments. Dysfunction or weakness in the core musculature can disrupt this balance, leading to altered movement patterns and impaired motor control. However, a significant gap persists in the literature regarding the investigation of the effects of core stability exercises on motor control impairment. While core stability exercises have demonstrated efficacy in addressing pain and disability outcomes, their specific impact on motor control impairment in patients with low back pain remains underexplored. This gap underscores the need for further research to elucidate the potential benefits of core stability exercises on motor control in this patient population.

ELIGIBILITY:
Inclusion Criteria:

* Both gender Presence of back pain for ≥6 weeks
* Age 30 -50 years
* MCI (Motor Control Impairment) complaints (pain provocation in static posture)
* Participants had 3 or more positive test out of six MCI tests.

Exclusion Criteria:

* LBP of specific cause, Recent spine surgery (<6 weeks)
* Comorbid health condition(Spondylolesthesis, fracture, Spondylolysis)
* Constant pain below knee
* Patient who denied consent

Ages: 30 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 44 (Actual)
Dates: Start 2024-09-01 (Actual); Primary Completion 2025-03-30 (Actual); Study Completion 2025-04-16 (Actual)

PRIMARY OUTCOMES:
MCI tests | baseline to 6 weeks
  First test is Waiters Bow test which includes flexion of hip 50-70⁰ in upright standing without movement (flexion) of low back. The second test is dorsal pelvic tilt in upright standing keeping thoracic spine neutral and lumbar spine moves towards flexion. The third tests involves normal standing to single leg stance and measurement of lateral movement of belly. Fourth test is upright sitting with knee extension. In this position lumbar spine should be neutral.
  Fifth test is quadruped position with pelvis moving back and fro i.e. rocking with low back in neutral. Hip should be flex 90-120⁰. The last test is prone lying with active knee flexion up to 90⁰ without movement of low back and pelvis. If 3 out 6 tests are positive then subject will be categorized as impaired motor control.

SECONDARY OUTCOMES:
NPRS | baseline to 6 weeks
  The NPRS is a self-reported, or clinician administered, measurement tool consisting of a numerical point scale with extreme anchors of 'no pain' to 'extreme pain'. The scale is typically set up on a horizontal or vertical line, ranges most commonly from 0-10 or 0-100, and can be administered in written or verbal form. The patient is asked to rate his/her pain intensity and a particular time frame or descriptor is established (e.g. within the last 24 hours, today, worst pain, average pain, or least pain
Oswestry Disability Index (ODI | baseline to 6 weeks
  The Oswestry Disability Index (aka the Oswestry Low Back Pain Disability Questionnaire) is an extremely important tool that researchers and disability evaluators use to measure a patient's permanent functional disability. There are 10 questions, for each question there is a possible 5 points; 0 for the first answer, 1 for the second answer, etc. Add up the total for the 10 questions and rate them on the scale at right. Indicating Mild, Moderate, Severe, Complete or No disability.

CONTACTS AND LOCATIONS:
Overall Officials: Aisha Razzaq, PHD*, Principal Investigator — Riphah International University
Locations (1):
- Rehman Medical Institute, Peshawar, Khybar Pakhtunkha, Pakistan

IPD SHARING:
Plan to Share IPD: No